CLINICAL TRIAL: NCT06081348
Title: A Randomized Placebo-Controlled Trial of Sertraline vs. Placebo in the Treatment of Anxiety in Children and AdoLescents With NeurodevelopMental Disorders
Brief Title: Sertraline vs. Placebo in the Treatment of Anxiety in Children and AdoLescents With NeurodevelopMental Disorders
Acronym: CALM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Azrieli Foundation (Funder) (Unknown); Canadian Institutes of Health Research (Funder) (Unknown); Ontario Brain Institute (Funder) (Unknown); McMaster University (Other); Western University (Other); Queen's University (Other); University of Alberta (Other); Alberta Health services (Other); St. Justine's Hospital (Other); Dalhousie University (Other); Unity Health Toronto (Other); University of Toronto (Other); The Hospital for Sick Children (Other); Maternal, Infant, Child and Youth Research Network (MICYRN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SER-11-2020
Record Dates: First submitted 2023-09-27; First posted 2023-10-13 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-11

CONDITIONS: Neurodevelopmental Disorders; Autism; Autism Spectrum Disorder; Fragile X Syndrome; Tuberous Sclerosis; 22Q11 Deletion Syndrome; 22Q11 Deletion; ADHD; Tic Disorders; Tourette Syndrome; Tourette Syndrome in Children; Tourette Syndrome in Adolescence; ADHD - Combined Type; ADHD Predominantly Inattentive Type; ADHD, Predominantly Hyperactive - Impulsive; Anxiety; Anxiety Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders; Autistic Disorder; Autism Spectrum Disorder; Fragile X Syndrome; Tuberous Sclerosis; 22q11 Deletion Syndrome; DiGeorge Syndrome; Attention Deficit Disorder with Hyperactivity; Tic Disorders; Tourette Syndrome; Anxiety Disorders | interventions — Sertraline; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sertraline (Active Comparator)
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sertraline — Oral capsule (25mg, 50mg, 100mg, 200mg)
  Other Names: Sertraline Hydrochloride; Zoloft; Serotonin Reuptake Inhibitor
  Arms: Sertraline
Other: Placebo — Oral placebo capsule
  Arms: Placebo

SUMMARY:
There are currently no approved medications for the treatment of anxiety in children and youth with neurodevelopmental disorders (NDDs), both common and rare. Sertraline, a selective serotonin reuptake inhibitor, has extensive evidence to support its use in children's and youth with anxiety but not within NDDs. More research is needed to confirm whether or not sertraline could help improve anxiety in children and youth with common and rare neurodevelopmental conditions. This is a pilot study, in which we plan to estimate the effect size of reduction in anxiety of sertraline vs. placebo. across rare and common neurodevelopmental disorders, and determine the best measure(s) to be used as a primary transdiagnostic outcome measure of anxiety, as well as diagnosis specific measures in future, larger-scale clinical trials of anxiety in NDDs.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients 8-17 years of age, inclusive
2. Females of child bearing potential who are sexually active and agree to use medically acceptable birth control throughout the study and at least one week post last dose of study drug.
3. Meet Diagnostic and Statistical Manual of Mental Disorders - DSM-5 criteria for ASD, ADHD, Tic Disorders, or genetic diagnosis of Fragile X, tuberous sclerosis or 22q11 deletions.
4. Meet DSM-5 criteria for one of the following anxiety disorders: Separation Anxiety Disorder, Social Anxiety Disorder, Agoraphobia, Generalized Anxiety Disorder, or Unspecified Anxiety Disorder, based on expert clinical interview, supported by the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS; Kaufman et al., 2016). Other specified anxiety disorder is included to account for youth with impairing anxiety symptoms who may not meet criteria for one of the other anxiety disorders.
5. Have a Clinician's Global Impression-Severity for anxiety (CGI-S; Guy, 1976)) score ≥ 4 (moderately ill) (inter-rater reliability will be done prior to initiation of enrollment, using videotapes of interviews and vignettes)
6. Have at least phrase speech, to allow for some self-report. So that results can be generalized to children and youth with NDD and various levels of ability, no IQ cut-off will be employed. Full-scale IQ (as measured by the Stanford-Binet) is measured to explore its effect on efficacy and safety*
7. If already receiving interventions, must meet the following criteria:

   1. If receiving concomitant medications affecting behaviour, must be on a stable dose during the month prior to screening and will not electively modify ongoing medications for study duration
   2. If already receiving stable non-pharmacological behavioural interventions, have stable participation during 3 months prior to screening, and will not electively modify ongoing interventions
8. Ability to complete assessments in English/French

Exclusion Criteria:

1. Receiving other SSRIs within four weeks of randomization (6 weeks for fluoxetine)
2. Previous treatment with sertraline, at an adequate dose (at least 100mg for 6 weeks, or lower dose and duration if not well-tolerated), associated with no response or significant-to-the-participant side effects.
3. Received more than 2 previous appropriate trials of SSRIs with no adequate response
4. Pregnant females or sexually active females on inadequate contraception
5. Serious medical condition that, based on Investigator judgment, might interfere with the conduct of the study, confound interpretation of the study results, or endanger participant. In addition diabetic patients on medications for glycemic control will be excluded as sertraline may interfere with glycemic control.
6. Hypersensitivity to sertraline or any components of its formulation
7. On Monoamine Oxidase Inhibitors or pimozide (as per product monograph)
8. On concomitant medications known to significantly increase QT interval where this would result in unacceptable risk per Investigator judgment.
9. Known congenital QT prolongation
10. HIV, hepatitis B or C, hemophilia, abnormal blood pressure, substance abuse, immunity disorder, major depressive episode or psychosis (as required by Health Canada)
11. Unable to tolerate venipuncture
12. Unable to swallow capsules
13. Enrolled in another intervention study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The Screen for Child Anxiety Related Emotional Disorders (SCARED) - parent version | 16 weeks
  The SCARED is a 41-item measure of anxiety symptoms, with both child and parent versions. The parent version will be used as a primary outcome measure. The minimum overall score is 0 while the maximum overall score is 82. A score greater than or equal to 25 may indicate the presence of an Anxiety Disorder. Higher scores indicate a higher instance of anxiety symptoms while a lower score indicates a lower instance of anxiety symptoms.

SECONDARY OUTCOMES:
Clinical Global Impressions - Improvement Scale - Global (CGI-I) | 16 weeks
  The CGI-I is a clinician reported scale which will be used to examine the effect of sertraline vs. placebo on measures of global function. The CGI-Improvement Scale employs a seven point (1 = very much improved to 7 = very much worse) to determine the participant's improvement in response to treatment.
Adverse events | 16 weeks
  Adverse events as elicited by the SMURF.
Pediatric Quality of Life Inventory (PedsQL) | 16 weeks
  The PedsQL will be used to examine the effect of sertraline vs. placebo on measures of quality of life. The PedsQL is measuring health-related quality of life (HRQOL) in 2- to 18-year-olds. The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent-proxy report scales that have been used extensively as an outcome measure, including in ASD. We will use the parent-proxy report scale, and optionally, age-appropriate child self-report scale. Each item is is rated between a 0 (Never a problem) to 4 (Almost always a problem).
Whole blood serotonin (5-HT) assessment | 16 weeks
  A whole blood serotonin assessment will be completed to examine the effect of sertraline vs. placebo on biomarkers of serotonin. 3mL of blood will be drawn at screening and week 16 visits for the purpose of this assessment. High performance liquid chromatography will be performed using fluorometric detection of 5-HT, tryptophan (TRP), and 5-hydroxyindole acetic acid (5-HIAA), using N-methylserotonin as an internal standard. Using this method, 5-HT intra- and inter- assay coefficients of variation are reliably less than 5% and 10%, respectively.
Clinical Global Impressions- Improvement Scale (CGI-I) focused on anxiety | 16 weeks
  The CGI-I is a clinician reported scale which will be used to examine the effect of sertraline vs. placebo on measures of global anxiety. The CGI-Improvement Scale employs a seven point (1 = very much improved to 7 = very much worse) to determine the participant's improvement in response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Evdokia Anagnostou, Principal Investigator — Holland Bloorview Kids Rehab Hospital
Locations (8):
- Canada (8):
  - Alberta Children's Hospital - University of Calgary, Calgary, Alberta
  - University of Alberta-Glenrose, Edmonton, Alberta
  - Dalhousie University - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University of Western Ontario, Lawson Health Research Institute, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - Ste Justine Hospital - Universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Through Brain Code
URL: https://braininstitute.ca/